CLINICAL TRIAL: NCT07337122
Title: Postoperative Swallowing and Voice Outcomes After Collagen Matrix Reconstruction in Oral and Oropharyngeal Cancer Surgery
Brief Title: Collagen Matrix in Oral Cancer Surgery
Status: Completed | Type: Observational
Sponsor: SAYAH Charline (Other)
Responsible Party: Sponsor-Investigator, SAYAH Charline, Dr SAYAH Charline, Hôpital de la Croix-Rousse
Organization: Hôpital de la Croix-Rousse (Other)
Other Study IDs: 2020/104
Record Dates: First submitted 2025-12-21; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Oral Cancer , Oral Squamous Cell Carcinoma, Oral Cavity Cancer; Oropharynx Squamous Cell Carcinoma; Oropharynx Cancer
Keywords: oral cancer; phonation; swallowing; voice; glossectomy; reconstruction; tachosil
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case group: Patient were ≥18 years with a histologically confirmed squamous cell carcinoma or other malignant tumor of the oral cavity and/or oropharynx with surgical resection indicated (T1-T3). The performance status was betwen 0 and 2. Patients were receiving or not receiving postoperative adjuvant radiotherapy

SUMMARY:
This study tend to evaluate postoperative phonation and swallowing after oncologic surgery of the oral cavity or oropharynx with application of a collagen matrix (Tachosil®). Patients are asked to complete a questionnaire the day before the surgery and at 1 and 6 months after.

DETAILED DESCRIPTION:
It was an interventional study with a single Group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed squamous cell carcinoma or other malignant tumor of the oral cavity and/or oropharynx
* Performance status (PS) 0-2
* Tumor stages for which surgical resection was indicated (T1-T3)
* Patients receiving or not receiving postoperative adjuvant radiotherapy

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Inability or anticipated poor compliance with study procedures
* Missing questionnaire data
* Congenital or acquired swallowing disorders (neurological or neuromuscular disease)
* Congenital or acquired speech disorders (neurological or neuromuscular disease)
* Death during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were selected among patients presenting to the ENT department of the University Hospital of Besançon for a suspected lesion of the oral cavity or oropharynx.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Swallowing evaluation | From enrollment (the day before the surgery) to 6 months postoperatively.
  We use the Deglutition Handicap Index questionnaire to evaluative swallowing before and after surgery. Patients completed the questionnaires the day before surgery, and at 1 month and 6 months postoperatively.
Voice evaluation | From enrollment (the day before the surgery) to 6 months postoperatively.
  We use the Voice Handicap Index questionnaire to evaluate the phonatione before and after surgery. Patients completed the questionnaires the day before surgery, and at 1 month and 6 months postoperatively.

SECONDARY OUTCOMES:
Length of hospital stay | From the day before the surgery up to 3 weeks after surgery. The number of days between hospital admission and discharge to home was calculated.
  We evaluate the length of hospital stay, it was expressed in days as mean and standard deviation
time to oral feeding resumption | From the surgery up to two weeks.
  Number of days between the surgery and the time the patient start to eat again by the mouth.
incidence and onset of device-related complications | From the day of the surgery to one week after
  Incidence of immunologic reaction to the collagen matrix (tachosil). Expressed in number and pourcentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitary Hospital of Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided